CLINICAL TRIAL: NCT05285865
Title: Effects of Scapular Mobilization on Inspiratory Capacity of Post-CABG Patients
Brief Title: Scapular Mobilization on Inspiratory Capacity of Post-CABG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01278 Sakina Asghar
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: CABG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Thrice a day ,Conventional treatment according to American Heart Association Guidelines i.e., Incentive spirometer, chest clearance, expectoration of the sputum (suctioning if needed), mobilizing the patient out of bed, AAROM and AROM exercises.
  Interventions: Other: Conventional Treatment
- Scapular Mobilization (Experimental): Thrice a day Scapular mobilization (SM) along with Conventional treatment
  Interventions: Other: Scapular Mobilization

INTERVENTIONS:
Other: Conventional Treatment — Thrice a day for complete length of stay. This is Conventional treatment The total duration of session will be of 15-20 mins.
  Arms: Conventional Treatment
Other: Scapular Mobilization — Thrice a day for complete length of stay including two sets of repetitions with a rest interval of 30 seconds between sets. Grade 1-3 As reported in a study Scapular mobilization (SM) i.e., Scapular superior, inferior glides, upward and downward rotations and scapular distraction, along with Conventional treatment according to American Heart Association Guidelines i.e., Incentive spirometer, chest clearance, expectoration of the sputum (suctioning if needed), mobilizing the patient out of bed, AAROM and AROM exercises.
  Arms: Scapular Mobilization

SUMMARY:
To determine the effects of scapular mobilization on pulmonary functions of post-CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* CAD patients undergone CABG surgery (Post-Op. Day#. 01).
* Both genders (male and female).
* Aged between 40 to 70 years .
* Patient having oxygen saturation (SPO2) of more than or equal to 90% with 25% of fraction of inspired oxygen (FiO2) - (possibly nasal cannula inserted).

Exclusion Criteria:

* Patients with low glasgow coma scale (GCS) score (less than 15).
* Patients having inspiratory capacity of 3500ml and above.
* Patients on ventilator.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incentive Spirometer | 1 week
  An incentive spirometer is a device that will expand the lungs by helping the patient breathe more deeply and fully
Borg scale | 1 week
  The Borg Rating of Perceived Exertion (RPE) is a way of measuring physical activity intensity level.
Numeric pain rating scale | 1 week
  What is a numerical pain rating scale? The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain
Digital Spirometer | 1 week
  Spirometer is a portable lung function testing device, which mainly used to examine lung function related parameters for patients

CONTACTS AND LOCATIONS:
Overall Officials: Malik Muhammad Ali Awan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No